CLINICAL TRIAL: NCT05657600
Title: Effectiveness of Video-based Yoga Practices on the Physical Features, Respiratory Capacity and Sleep Quality of Sedentary Women in Pandemic Days
Brief Title: Effectiveness of Video-based Yoga Practices for Sedentary Women in Pandemic Days
Acronym: YogaVideo
Status: Completed | Type: Observational
Sponsor: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Habibe Serap Inal, Prof.Dr, Istanbul Galata University
Other Study IDs: IstanbulGalataU
Record Dates: First submitted 2022-11-08; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Women
Keywords: video-based yoga; Posture; Vital capacity; Exercise; Fatigue
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Quality of Life; Sleep; Functional Status; Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Video-based yoga group: The pranayama (respiration), asana (poses), yoga exercises and meditation were given to by means of video at home for 6 weeks (2days/week) as 12 sessions, and 60 min.
  Interventions: Behavioral: Sociodemographic profile, quality of life, sleep, fatigue, physical function and balance assessments; Other: Video-based yoga
- Face-to-face yoga group: The pranayama (respiration), asana (poses), yoga exercises and meditation were given to face to face at Volunteer Training and Consultation Centre for 6 weeks (2days/week) as 12 sessions, and 60 min.
  Interventions: Behavioral: Sociodemographic profile, quality of life, sleep, fatigue, physical function and balance assessments; Other: Face-to-face yoga
- physical exercise: The exercises for respiration, muscle strengthening, stabilization, and flexibility were given face-to-face at Volunteer Training and Consultation Centre for 6 weeks (2days/week) as 12 sessions, and 60 min.
  Interventions: Behavioral: Sociodemographic profile, quality of life, sleep, fatigue, physical function and balance assessments; Other: physical exercise

INTERVENTIONS:
Behavioral: Sociodemographic profile, quality of life, sleep, fatigue, physical function and balance assessments — Respiratory functions are assessed with a portable spirometer according to the criteria of the American Thoracic Society and European Respiratory Society. Measures the physical, mental, social, and environmental well-being were tested to understand the quality of life. The quality of sleep, delayed sleep, sleep disorders, usage of sleeping pills, and loss of functionality during the day were assessed. The balance and static standing capability of the participants were tested. The functional reach of participants were tested by expecting them to lean forwardly as far as they can without taking a step, nor rising their heels. The fatigue feeling of the participants as everyday life were assessed. The posture of the participants was assessed on 13 regions at anterior, posterior and lateral views.
Other: Video-based yoga — Video-based yoga
  Groups: Video-based yoga group
Other: Face-to-face yoga — Face-to-face yoga
  Groups: Face-to-face yoga group
Other: physical exercise — physical exercise
  Groups: physical exercise

SUMMARY:
This is an observational study aiming to Examine the effects of video-based yoga compared to face-to-face yoga and physical exercise practices on the physical features, respiratory capacity and sleep quality of sedentary women in pandemic days.

The pranayama (respiration), asana (poses), and meditation were given to the face-to-face yoga group, and the same exercises of the face-to-face yoga group were recorded in the video for the video-based yoga group. The exercises for respiration, muscle strengthening, stabilization, and flexibility were given face-to-face to the physical exercise group.

DETAILED DESCRIPTION:
This is an observational study aiming to Examine the effects of video-based yoga compared to face-to-face yoga and physical exercise practices on the physical features, respiratory capacity and sleep quality of sedentary women in pandemic days.

The respiration, poses, and meditation were given to the face-to-face yoga group, and the same exercises of the face-to-face yoga group were recorded in the video for the video-based yoga group. The exercises for respiration, muscle strengthening, stabilization, and flexibility were given face-to-face to the physical exercise group. The sessions for each group were given for a total of 6 weeks (2days/week) as 12 sessions, and 60 min. Their respiration (spirometer Pony-Fx), sleep (Pittsburgh Sleep Quality Index), posture (New York Posture Rating Chart), balance (Single Leg Stance Assessment, Functional Reach Distance), functional strength (5X Sit-to-Stand test), fatigue (Fatigue Severity Scale) and quality of life (WHOQOL-BREF) were evaluated at the beginning and end of the 6 weeks. The data were assessed statistically.

ELIGIBILITY:
Inclusion Criteria:

* being between the age of 18 - 60 years,
* not having any history of a systemic disease, such as musculoskeletal or neurological problems, cardiac or lung diseases, diabetes and no history of recent surgery
* not having participated in a regular exercise program in the last 6 months and
* not having a history of active sports engagement

Exclusion Criteria:

* not being voluntary to join the study and
* missing more than three sessions during the study period

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sedentary women adults
Study Population: Sedentary adult women
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Tests | 2 months
  Respiratory Function (portable spirometer; Pony Fx, Rome, Italy) assessed according to the criteria of the American Thoracic Society and European Respiratory Society. The deep expiration after maximal inspiration aForced Vital capacity-FVC(lts), the air volume released in the first second during forced expiration - Forced Expiratory Volume 1-FEV1(lts), the ratio of forced expiratory volume to the forced vital capacity in the first second - FEV1/FVC (%), peak expiratory flow during forced expiration - PEF (lt/sec) and vital capacity - VC (lts) are evaluated.
The demographic data of the participants | 2 months
  The demographic data of the participants as gender, age, dominant hand, educational background, smoking status, and the number of cigarettes per day were recorded by means of a specially prepared questionnaire for this study.
body weight, height and body mass index of the participants | 3 months
  The body weight (kilograms), height (meters) will be measured and the body mass index (kg/m2) of each participant will be recorded.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index-PSQI | 2 months
  It is a self-reporting scale that is comprised of 19 items. Each element of the scale is evaluated on a score of 0 to 3 equally. Questions are assigned a score between 0 and 3 and higher scores reflect bad sleep quality.The total PSQI score (0-21) as scale is acquired after the addition of the sub scales in the questionnaire. High values indicate bad sleep quality and a higher level of sleep disturbance. A total score above 5 indicates that the quality of sleep is poor clinically.

OTHER OUTCOMES:
5X Sit-to-Stand test | 2 months
  It is a test to evaluate the functional strength of the lower extremities. The participants were asked to cross the arms on their chest while sitting on the chair and then stand up and sit on a chair as quickly and without stopping as possible, the elapsed time (minutes) at the end of the fifth repetition was recorded.
The Single-Leg Stance Test | 2 months
  It is a test to evaluate the balance and static standing capability of the participants. The participant was asked to lift one foot, while standing. The time ( minutes) was stopped, once the foot touch the floor
The Functional Reach test | 2 months
  It is a test to assess the functional reach of the participants. They were asked to stand by the wall at their dominant side with 90-degree shoulder flexion, 180-degree elbow extension, and with a closed fist; keep their feet apart from each other at their hip-width. The level of the head of the 3rd metacarpal bone was marked over the ruler horizontally attached to the wallis marked. Then, the participant was asked to "lean forwardly as far as they can without taking a step, nor rising their heels". The place where the 3rd metacarpal head of the participants reached was marked again. After three trials the amount of reaching (cm) that was the distance between the initial and the final mark was measured and the average was recorded.
Fatigue Severity Scale | 2 months
  It was used to measure the fatigue feeling of the participants as everyday life. Each item of the scale was comprised of 7 scorings with 9 items in total. The arithmetic average of the total score was taken. Cases with a score of 4 and above were considered in the fatigue group.
New York Posture Assessment Test | 2 months
  It is used to assess the posture from anterior, posterior and lateral sides as A-head, B- shoulder levels, C- spine, D- hip levels, E- feet; and mediolaterally, F-feet arches; and at posterior side: G- head, H-chest, I-shoulders, J- upper, K- trunk, L- abdomen, M- low back. They were scored as (5) for good-normal, (3) for moderately affected, (1) severely affected postures. The score is between 65-13 with the cut-off score ≥ 45 is very good, 44-40 is good, 39-30 is moderate, 29-20 is poor, ≤ 19 is bad posture.
The World Health Organization Quality of Life-BREFF | 2 months
  The questionnaire assessing the quality of life of the participants consists of 26 questions and measures of physical, mental, social, and environmental well-being adult population were assessed. The Turkish version has 27 questions the 27th was named the Environment-Turkish. The area scores are calculated between 1 and 100. As the scores increase, the quality of life increases as well.
  It is a self-reporting scale that is comprised of 19 items. Each element of the scale is evaluated on a score of 0 to 3 equally. Questions are assigned a score between 0 and 3 and higher scores reflect bad sleep quality.The total PSQI score of 0-21 is acquired after the addition of the sub scales. High values indicate bad sleep quality and a higher level of sleep disturbance. A total score above 5 indicates that the quality of sleep is poor clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap İnal, PhD, Study Director — Istanbul Galata University; Nahide Kocer, MSc, Principal Investigator — Dogus Universitesi
Locations (1):
- Kadıkoy Municipality Rasimpasa Volunteer Training and Consultation Centre, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No